CLINICAL TRIAL: NCT07130591
Title: Investigation of the Efficiency of the Cogniplat Gaming Platform on Cognitive Functions in Geriatric Individuals: a Randomized Controlled Trial
Brief Title: Efficiency of CogniPlat on Cognitive Functions in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: cogniplat
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: cogniplat; geriatric rehabilitation; cognitive games
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This prospective, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Play Group (Experimental): Group of patients treated with the Cogniplat gaming platform
  Interventions: Other: Cogniplat game platform
- Control Group (Other): Individuals in this group did not participate in any regular play program
  Interventions: Other: Control group

INTERVENTIONS:
Other: Cogniplat game platform — The Cogniplat gaming platform is designed to improve cognitive function in geriatric individuals, with or without mild cognitive impairment. Participants played the Cogniplat games face-to-face with a physiotherapist twice a week on non-consecutive days for 10 weeks, sessions lasting about 30-45 minutes. Scores from the platform were recorded to evaluate progress.
  Other Names: CGP
  Arms: Play Group
Other: Control group — Individuals in this group did not participate in any regular play program. Demographic data were recorded. For evaluation purposes, a single session of Cogniplat game platform was applied in the first interview and in the second interview 10 weeks later. Initial and final evaluations were recorded.
  Other Names: CG
  Arms: Control Group

SUMMARY:
Mild cognitive impairment is a common intermediate stage between normal aging and dementia, affecting memory and other cognitive domains in older adults. While pharmacologic treatments lack strong evidence, exercise, cognitive training, and game-based interventions have shown positive effects on cognitive functions. The Cogniplat gaming platform, designed to improve cognitive abilities through personalized, multidisciplinary game exercises, has not yet been clinically evaluated. The present study aims to assess the effectiveness of Cogniplat in enhancing cognitive functions in geriatric individuals.

DETAILED DESCRIPTION:
Mild cognitive impairment may occur with physiological aging in geriatric individuals. This describes an intermediate stage from normal cognitive status to dementia. In mild cognitive impairment, there is cognitive impairment in both memory and non-memory domains. Anxiety, depression and other adverse mental health conditions also lead to decreased cognitive functioning. The risk of mild cognitive impairment turning into dementia is quite high. Therefore, diagnosis, follow-up and treatment are important issues. Mild cognitive impairment is common in geriatric populations. Its prevalence increases with age and low education level. The incidence of mild cognitive impairment in geriatric individuals aged 65 years and older is 15-20%.

There is no high quality evidence showing the efficacy of pharmacologic agents in the treatment of mild cognitive impairment. There are also studies showing that exercise and cognitive training have an improving effect on cognitive functions. Cognitive games also have a stimulating effect on memory and communication in these individuals. Game-based education reduces the risk of mild cognitive impairment and depression by stimulating the cerebral cortex and also motivates older adults to participate in treatment. Computer-based cognitive gaming training has been found to have positive effects on attention ability and memory development in this population.

The Cogniplat game platform used in the study is a rehabilitation tool developed to improve the cognitive functions of elderly individuals. Cogniplat is based on a multidisciplinary approach combining theories from neuropsychology, cognitive linguistics and speech therapy. It focuses on improving cognitive functions through different game exercises. In addition, Cogniplat automatically adjusts the difficulty and type of exercises by detecting the cognitive needs of individuals. In the literature, the Cogniplat game platform has been developed, but no studies evaluating its effectiveness have been found. Therefore, the present study was planned to examine the effect of the "Cogniplat" game platform on cognitive functions in geriatric individuals.

ELIGIBILITY:
Inclusion Criteria:

* To volunteer to participate in the study
* To be over 65 years old
* had a mini-mental test score above 24
* could use smartphones and tablets
* To have sufficient reading and writing skills to use the gaming platform
* To have good cooperation skills and not have a disease causing vision loss

Exclusion Criteria:

* Individuals with orthopedic or neurological conditions that prevent the use of a tablet with the upper extremities
* Individuals who are unable to maintain sitting balance
* Individuals with hearing loss that may prevent them from hearing information related to the gaming platform

Ages: 65 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Mini-Mental Test | At baseline and 10 week after
  The Mini-Mental Test consists of eleven items under five main headings: orientation, recording memory, attention and calculation, recall and language, and is evaluated on a total of 30 points. A score of 23/24 is accepted as the threshold for the diagnosis of mild dementia in Turkish elderly
Game Platform Scoring | At baseline and 10 week after
  For each game played on the platform, game duration, accuracy and speed variables were recorded on the servers connected to the platform. Individuals in both the study and control groups played a game on the platform, and the score of this game was recorded on the system and used in the analysis.Game duration, accuracy and speed will be aggregated into a single game performance score automatically generated by the platform and recorded for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Betül Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University; Ayşe Sezgi Kızılırmak Karataş, Pt.PhD, Principal Investigator — Izmir Democracy University; Nuri Üçler, Msc.Pt., Principal Investigator — Ege University; Ebru Köse, Pt.PhD, Principal Investigator — Izmir Democracy University; Cansu Ozdemir, Msc.Pt, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy Univercity, Izmir, Turkey (Türkiye)